CLINICAL TRIAL: NCT00900120
Title: Banking DNA for Analysis of Genetic Polymorphisms in Patients With Cancer
Brief Title: Collecting and Storing Blood Samples From Patients With Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Will be replaced by honest broker program
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0220044856; P30CA072720 (NIH); CINJ-000402; CINJ-IRB-4856
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Nonmalignant Neoplasm; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: aplastic anemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; secondary myelodysplastic syndromes; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage 0 chronic lymphocytic leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated hairy cell leukemia; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage II childhood lymphoblastic lymphoma; stage II childhood small noncleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; Burkitt lymphoma; childhood diffuse large cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood immunoblastic large cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; childhood myelodysplastic syndromes; recurrent childhood anaplastic large cell lymphoma; stage I childhood anaplastic large cell lymphoma; stage II childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neoplasms; Anemia, Aplastic; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Recurrence; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Dendritic Cell Sarcoma, Interdigitating; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Collecting and storing samples of blood from patients with cancer to test in the laboratory may help the study of cancer in the future.

PURPOSE: This research study is collecting and storing blood samples from patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish a repository for long-term storage of DNA obtained from patients treated at the Cancer Institute of New Jersey.
* To establish a mechanism whereby investigators can analyze correlations between genetic polymorphisms and clinical outcomes (e.g., response to treatment).

OUTLINE: Additional blood samples are collected for banking from patients while they are scheduled for routine blood draw as a part of their normal care. Samples are stored in a secure place under the control of the Cancer Institute of New Jersey Tissue Retrieval service. The samples may be used for DNA, RNA, or protein extraction and analyses, as well as generation of cell lines.

Demographic data (ethnicity, race, age, and sex), diagnosis, family history, and previous treatments (chemotherapy, radiation, and surgery) are recorded on the case report form and kept in a secure location in the Office of Human Research Services (OHRS).

Patients may have their samples removed and destroyed at any time.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy or bone marrow disorder (i.e., myelodysplasia, myeloproliferative syndrome, or aplastic anemia)
* Must be undergoing treatment or planning to undergo treatment at the Cancer Institute of New Jersey

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen at CINJ who have a diagnosis of cancer and plan to be treated at CINJ will be asked to participate in this DNA banking resource
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
DNA repository for long-term storage of DNA obtained from patients treated at the Cancer Institute of New Jersey | Indefinite
Investigative mechanism to allow correlations between genetic polymorphisms and clinical outcomes | Indefinite

CONTACTS AND LOCATIONS:
Overall Officials: Kim Hirshfield, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey